CLINICAL TRIAL: NCT03380104
Title: Intradural Percutaneous Stimulation - Inducing Physiological Responses.
Brief Title: Intradural Percutaneous Stimulation
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to obtain FDA IDE approval. Currently working on additional preclinical testing.
Sponsor: Matthew Howard (Other)
Responsible Party: Sponsor-Investigator, Matthew Howard, MD, Professor and Chairman, University of Iowa
Organization: University of Iowa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 201708754
Record Dates: First submitted 2017-10-24; First posted 2017-12-20 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Pain, Chronic
Keywords: Percutaneous Electrical Nerve Stimulation
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Intervention Model Description: All subjects enrolled in this study will undergo Intradural Spinal Cord Stimulation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Single Arm (Experimental): Intradural Spinal Cord Stimulation; Administration of Questionnaires
  Interventions: Device: Intradural Spinal Cord Stimulation; Behavioral: Administration of Questionnaires

INTERVENTIONS:
Device: Intradural Spinal Cord Stimulation — The device will be placed percutaneously at the lumbar spine at L2-3 or L3-4 level into the intrathecal CSF space and advanced to the T8-10 disc space. After positioning of the intrathecal lead, the stimulation catheter will be run through a standardized experimental algorithm consisting on various frequencies.
Behavioral: Administration of Questionnaires — Subjects will be administered questionnaires to evaluate pain, quality of life, and global function prior the study, at 1 hour after the completion of the study, and at 4 day follow-up appointment.

SUMMARY:
The purpose of the study is to test the effects of intradural, spinal cord stimulation using a device placed in the same manner as a lumbar drain performed during a standard epidural spinal cord stimulation (SCS) trial routinely performed prior permanent lead and stimulation device implantation.

DETAILED DESCRIPTION:
In this pilot study the investigators will test an ability of intradural electrical stimulation in humans to elicit physiological responses (paresthesia or tingling sensation) and decrease pain when placed in the region of the thoracic spinal cord in a controlled manner. This subject population is comprised of patients that had previously failed various conservative pain management treatment plans and are deemed candidates for treatment of pain by spinal cord stimulation. The investigators will use commercially available device to deliver an intradural electrical stimulation to the spinal cord. This device is FDA approved for intracranial electrophysiological monitoring and delivery of electrical stimulation of the subsurface level of the brain.

As a part of the study, the subject will be offered to complete the following questionnaires to assess quality of life and global function. These questionnaires will be completed prior the procedure and at specified time periods following the research intervention. The experimental portion of the procedure will follow the standard epidural spinal cord stimulator testing. Under fluoroscopic guidance, using a paramedian approach and shallow entry angle, the device will be placed percutaneously at the lumbar spine at L2-3 or L3-4 level into the intrathecal cerebrospinal fluid (CSF) space and advanced to the T8-10 disc space. The stimulation catheter will run through a standardized experimental algorithm further described in greater details. The initial stimulation will last approximately 30 minutes and involve testing for paresthesias (tingling) and measurement of the threshold signal strength for onset of this sensation at 60 hertz (Hz) and 10000 Hz frequences. During this portion the subject will be asked to describe the sensations and rate his or her pain on a 0 to 10 scale. Following this initial stimulation, the frequency will be changed to 10 kilohertz (KHz) to run over the period of 4 hours. The investigators will continue evaluating the effects of stimulation using visual analogue scores during this period of time.

ELIGIBILITY:
Inclusion Criteria:

* Patients with neuropathic pain and concordant neurological findings previously consented for an epidural spinal cord stimulator trial
* Patients greater than 18 years of agree
* Must have one of the following:

  1. Diagnosed with medically refractory chronic neuropathic pain, post laminectomy pain syndrome, or failed back surgery syndrome and planning to undergo a spinal cord stimulation trial
  2. Been deemed refractory to all other treatments and would otherwise receive an intrathecal catheter/pump for chronic narcotic administration
* Disease duration of at least 6 months with no lasting success with standard therapies or medications with exception of spinal cord stimulation
* Mean pain intensity of a least 5 (or greater) measured on a visual analogue scale from 0 (no pain) to 10 (severe pain)
* MRI or CT Myelogram of the lumbar and thoracic spine (within 12 months prior to screening)
* No compressive spinal pathology or intradural implants (eg., syrinx shunt tubes)
* Psychological screening has been completed and the patient has been cleared by a psychologist or psychiatrist as a suitable SCS candidate
* Female patients of childbearing potential must have a negative serum pregnancy test
* Patients agree to comply with the study protocol and have reviewed and given written informed consent

Exclusion Criteria:

* Patients who are unable or unwilling to provide feedback regarding the response
* Subject has an existing intrathecal drug pump
* Pain is attributed to: vascular disorder; musculoskeletal disorder; substance abuse or withdrawal; infection; disorder of homeostasis
* Subject is currently enrolled in another trial
* History of coagulation disorders or patients on chronic anticoagulant or antiplatelet therapy that is not able to be safely held for 14 days
* History of thoracic trauma or spinal surgery extending into the thoracic spine
* History of arachnoiditis or intradural spinal surgery that would limit catheter insertion to the target site
* Current clinically significant or disabling chronic pain problem or condition that is likely to confound evaluation of the study endpoints (i.e. chronic migraine, significant arthritis of the hip associated with primary groin pain complaint)
* Radiographic evidence of frank spinal instability (gross mobile spondylolisthesis or abnormal subluxation requiring fusion, calcific arachnoiditis, or severe thoracic or lumbar stenosis
* Subject has a condition that requires diathermy or repeated MRIs
* New medication for pain initiated within 8 weeks prior to initial baseline research evaluation
* Life expectancy less than 3 months
* Systemic infection or local infection of the spine or skin in the anticipated region of catheter insertion.
* Immune deficiency or history of post surgical infection
* Female candidates of childbearing potential who are pregnant (confirmed with a positive serum pregnancy test), not using adequate contraception as determined by the investigator, or nursing (lactating) a child
* Untreated or active psychiatric condition
* Complex regional pain syndrome or other condition that could limit testing or aggravate an ongoing medical condition
* Unresolved issues of secondary gain (i.e. litigation)
* The investigator deems that the subject is not suitable for the study even if they meet all other inclusive/exclusion criteria

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2020-06-01 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
Establishment of paresthesia threshold | 30 minutes
  Observe and record how various stimulation measures induce paresthesias and record this paresthesia threshold. This will be measured by having the patient state when they feel paresthesias as the stimulation amplitude is increased. This will be recorded as a raw number.
Establishment of motor threshold | 30 minutes
  Observe and record how various stimulation measures induce motor activity and record this motor threshold. This will be measured by having the patient state when they feel motor movement as the stimulation amplitude is increased. This will be recorded as a raw number.
Acute Adverse Pain Responses using short-form McGill Pain Questionnaire | 5 hours
  Demonstrate that intradural stimulation does not induce adverse painful responses during acute stimulation. Participants will be administered the short-form McGill Pain Questionnaire prior to start of testing and one hour following testing has concluded. The McGill Pain Questionnaire has a range of scores from zero (min) to 45(max) with lower numbers being better.
Acute Adverse Pain Responses using long form Brief pain inventory (BPI) | 5 hours
  Demonstrate that intradural stimulation does not induce adverse painful responses during acute stimulation. Participants will be administered the long form BPI prior to start of testing and one hour following testing has concluded. The brief pain index creates a severity and interference score that ranges from zero (min) and 10 (max) with lower numbers being better.

SECONDARY OUTCOMES:
Difference in Stimulation Intensity to induce paresthesias | 90 minutes
  Record the threshold difference in stimulation intensity between epidural and intrathecal stimulation. This will take the data collected from the patient's clinical epidural trial (paresthesia threshold) and compared to the patient's intradural threshold testing.
Unexpected/Chronic effects of stimulation | 1 month
  Record unexpected or unanticipated effects of stimulation that may limit its utility or conceivably provide a new avenue for neuromodulation not achievable with epidural stimulation. Participants will be contacted via telephone interviewed to screen for any unexpected outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew A Howard, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Charghi R, Chan SY, Kardash KJ, Finlayson RJ, Tran DQ. Electrical stimulation of the epidural space using a catheter with a removable stylet. Reg Anesth Pain Med. 2007 Mar-Apr;32(2):152-6. doi: 10.1016/j.rapm.2006.10.006. PMID 17350527
- [Background] Crews JC, Chan VWS. Perioperative management of patients and equipment selection for neural blockade. In: Cousins MJ, Horlocker TT, Bridenbaugh PO, Carr DB, Eds., Neural Blockade in Clinical Anesthesia and Pain Medicine (Wolters Kluwer, Philadelphia, 2009), Chap. 8, 160-180. ISBN-13: 978-0-7817-7388-1
- [Background] Flouty O, Oya H, Kawasaki H, Wilson S, Reddy CG, Jeffery ND, Brennan TJ, Gibson-Corley KN, Utz M, Gillies GT, Howard MA 3rd. A new device concept for directly modulating spinal cord pathways: initial in vivo experimental results. Physiol Meas. 2012 Dec;33(12):2003-15. doi: 10.1088/0967-3334/33/12/2003. Epub 2012 Nov 15. PMID 23151433
- [Background] Gibson-Corley KN, Flouty O, Oya H, Gillies GT, Howard MA. Postsurgical pathologies associated with intradural electrical stimulation in the central nervous system: design implications for a new clinical device. Biomed Res Int. 2014;2014:989175. doi: 10.1155/2014/989175. Epub 2014 Apr 1. PMID 24800260
- [Background] Howell B, Lad SP, Grill WM. Evaluation of intradural stimulation efficiency and selectivity in a computational model of spinal cord stimulation. PLoS One. 2014 Dec 23;9(12):e114938. doi: 10.1371/journal.pone.0114938. eCollection 2014. PMID 25536035
- [Background] Lena P, Martin R. Subdural placement of an epidural catheter detected by nerve stimulation. Can J Anaesth. 2005 Jun-Jul;52(6):618-21. doi: 10.1007/BF03015772. PMID 15983148
- [Background] Pope JE, Stanton-Hicks M. Accidental subdural spinal cord stimulator lead placement and stimulation. Neuromodulation. 2011 Jan;14(1):30-2; discussion 33. doi: 10.1111/j.1525-1403.2010.00299.x. Epub 2010 Oct 7. PMID 21992159
- [Background] Reddy CG, Dalm BD, Flouty OE, Gillies GT, Howard MA 3rd, Brennan TJ. Comparison of Conventional and Kilohertz Frequency Epidural Stimulation in Patients Undergoing Trialing for Spinal Cord Stimulation: Clinical Considerations. World Neurosurg. 2016 Apr;88:586-591. doi: 10.1016/j.wneu.2015.10.088. Epub 2015 Nov 14. PMID 26585728
- [Background] Sharpe AN, Jackson A. Upper-limb muscle responses to epidural, subdural and intraspinal stimulation of the cervical spinal cord. J Neural Eng. 2014 Feb;11(1):016005. doi: 10.1088/1741-2560/11/1/016005. PMID 24654267
- [Background] Toma AK, Papadopoulos MC, Stapleton S, Kitchen ND, Watkins LD. Systematic review of the outcome of shunt surgery in idiopathic normal-pressure hydrocephalus. Acta Neurochir (Wien). 2013 Oct;155(10):1977-80. doi: 10.1007/s00701-013-1835-5. Epub 2013 Aug 23. PMID 23975646
- [Background] Tsui BC, Gupta S, Finucane B. Detection of subarachnoid and intravascular epidural catheter placement. Can J Anaesth. 1999 Jul;46(7):675-8. doi: 10.1007/BF03013957. PMID 10442964
- [Background] Williams MA, Malm J. Diagnosis and Treatment of Idiopathic Normal Pressure Hydrocephalus. Continuum (Minneap Minn). 2016 Apr;22(2 Dementia):579-99. doi: 10.1212/CON.0000000000000305. PMID 27042909